CLINICAL TRIAL: NCT00655980
Title: Pharmacogenetics of Adverse Outcomes After Nitrous Oxide Anesthesia
Brief Title: Vitamins in Nitrous Oxide Study
Acronym: VINO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Foundation for Anesthesia Education and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: HSC 07-0592
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Major Surgery; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Vitamin B 12; Folic Acid; Nitrous Oxide; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment (Experimental): Vitamin B12 and folic acid
  Interventions: Drug: Vitamin B12 and folic acid
- Comparator (Placebo Comparator): Nitrous oxide and placebo
  Interventions: Drug: Nitrous oxide and placebo
- Standard of care (Other): standard of care
  Interventions: Other: standard of care

INTERVENTIONS:
Drug: Vitamin B12 and folic acid — 1 mg vitamin B12 IV 5 mg folic acid IV in 100 ml NS infusion
  Arms: Treatment
Drug: Nitrous oxide and placebo
  Arms: Comparator
Other: standard of care
  Arms: Standard of care

SUMMARY:
In this study, we want to find out if laughing gas (nitrous oxide) leads to a higher rate of cardiac complications after surgery in patients with a specific genetic profile (mutations in the MTHFR gene) and if this risk can be prevented by giving patients vitamin B12 and folate during surgery.

DETAILED DESCRIPTION:
Background and significance: Recent studies have shown that nitrous oxide (N2O) anesthesia may be associated with an increased risk of adverse cardiovascular outcomes. It is well-known that N2O inhibits vitamin B12-dependent enzymes and as a result increases plasma homocysteine concentrations. Homocysteine has been identified as risk factor for cardiovascular disease. Therefore elevations in homocysteine after N2O may be a causative factor in N2O toxicity. In a previous investigation, we found that patients who carry a homozygous mutation in the MTHFR gene develop higher homocysteine levels after N2O anesthesia than non-carriers. These patients might be at higher risk for adverse cardiac outcomes from N2O. Thus, there may be a pharmacogenetic mechanism to account for the adverse cardiac outcomes from N2O. Moreover, prevention of N2O-increased homocysteine concentrations in these high risk patients by perioperative vitamin B12 and folate supplementation might decrease the incidence of adverse cardiac outcomes.

Hypothesis: Patients carrying a homozygous MTHFR 677C>T or 1298 A>C variant allele will have a higher incidence rate of postoperative myocardial ischemia after N2O anesthesia [detected by serial TnI measurements] due to elevated homocysteine levels than normal "wild-type" non-carriers, and that the incidence rate will be reduced if they receive perioperative vitamin B12/folate supplementation.

Primary outcome: Myocardial ischemia in the first 72 hours after surgery (measured by serial troponin and ECGs).

Secondary outcome: Composite endpoint of 30-day mortality and major cardiac morbidity (non-fatal MI)

Design: Randomized controlled trial. 500 patients will receive N2O during surgery and will be randomized to receive B-vitamins or placebo. 125 patients will receive no N2O and no B-vitamins (control arm). Mendelian randomization of MTHFR genotype.

Intervention: IV vitamin B12 (1 mg) and folate (5 mg) pre- and postoperatively

Study setting: Barnes-Jewish-Hospital, St. Louis, MO

Patients: Patients scheduled for major surgery with or at risk for coronary artery disease

ELIGIBILITY:
Inclusion Criteria:

* Adult patients; age >18 yrs, ASA III-IV
* Previously diagnosed coronary artery disease or at risk for coronary artery disease
* Scheduled for major surgery (>2 hrs)

Exclusion Criteria:

* Patients not expected to live past 24 hours (ASA 5)
* Patients with significant pulmonary disease requiring supplemental oxygen
* Patients taking supplemental vitamin B12 or folate
* Contraindication against N2O (pneumothorax, mechanical bowel obstruction, middle ear occlusion, laparoscopic surgery, raised intracranial pressure)
* Hypersensitivity to cobalamins
* Leber's disease (hereditary optic nerve atrophy) [vitamin B12 interaction]
* Seizure disorder [folate interference]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 687 (Actual)
Dates: Start 2008-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Nagele, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 687 patients signed consent for enrollment; only 625 were analyzed.
Period: Overall Study
Arm/Group | Treatment | Comparator | Standard of Care
Started | 276 | 281 | 130
Completed | 250 | 250 | 125
Not Completed | 26 | 31 | 5
Not completed — surgery canceled; or subject or anesthes | 26 | 31 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Comparator | Standard of Care | Total
Number analyzed (Participants) | 250 | 250 | 125 | 625
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.6) | 65.2 (10.7) | 67.6 (10.9) | 65.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 97 | 45 | 234
  Male | 158 | 153 | 80 | 391
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 250 | 250 | 125 | 625
Smoking history [Count of Participants; unit: Participants] | 195 | 175 | 94 | 464
Diabetes [Count of Participants; unit: Participants] | 96 | 88 | 39 | 223
Hypertension [Count of Participants; unit: Participants] | 200 | 204 | 100 | 504
Chronic renal failute [Count of Participants; unit: Participants] | 16 | 35 | 16 | 67
on hemodialysis [Count of Participants; unit: Participants] | 1 | 3 | 1 | 5
Coronary artery disease [Count of Participants; unit: Participants] | 140 | 148 | 84 | 372
Congestive heart failure [Count of Participants; unit: Participants] | 27 | 31 | 15 | 73
Peripheral vascular disease [Count of Participants; unit: Participants] | 81 | 85 | 44 | 210
ASA staging [Count of Participants; unit: Participants] — ASA (American Society of Anesthesiologists) Physical status classification:
  ASA 1 = Normal healthy patient ASA 2 = Patient w/ mild systemic disease ASA 3 = Patient w/ severe systemic disease ASA 4 = Patient w/ severe systemic disease that is a constant threat to life ASA 5 = Moribund patient who's not expected to survive without the operation ASA 6 = Declared brain-dead patient, organs are being removed for donor purposes
  Higher values reflect worse disease status.
  Participants
    ASA 1-A normal healthy patient | 1 | 0 | 0 | 1
    ASA 2 A patient with mild systemic disease | 45 | 42 | 11 | 98
    ASA 3 - A patient with severe systemic disease | 199 | 196 | 106 | 501
    ASA 4 -A patient with severe systemic disease tha | 5 | 10 | 8 | 23
Lee's revised cardiac risk index (Mean [Mean (Standard Deviation); unit: units on a scale] — Lee's Revised Cardiac Risk Index Rapid pre-op assessment using the Revised Cardiac Risk Index
  Patients receive 1 point for meeting a criteria; then totaled to get their prospective risk level.
  High risk surgery Having Coronary Artery Disease Having Congestive Heart Failure Having Cerebrovascular Disease Having Diabetes Mellitus and on insulin Having a Serum Creatinine >2 mg/dl or >177 μmol/L
  Higher totals connote higher risk (range 0-6)
  units on a scale | 1.9 (0.8) | 2.0 (0.9) | 2.1 (0.8) | 2.0 (0.8)
Plasma total homocysteine mol/L [Mean (Standard Deviation); unit: mcmol/L] | 13.5 (5.7) | 13.4 (5.8) | 11.6 (4.2) | 13.1 (5.5)
MTHFR C677T polymorphism [Count of Participants; unit: Participants] — The MTHFR C677T polymorphism reduces MTHFR enzyme activity; therefore, these patients have higher risk factors for coronary artery disease, acute myocardial infarction, peripheral vascular artery disease, stroke, or venous thromboembolism; having increased basal homocysteine levels or an abnormal methionine-load test (e.g., deficiency of vitamins B12, B6, and folic acid). Population: Some patients had missing genotype
  Participants
    number analyzed (Participants) | 242 | 245 | 102 | 589
    677CC | 137 | 130 | 57 | 324
    677CT | 76 | 89 | 37 | 202
    677TT | 29 | 26 | 8 | 63
MTHFR A1298C plymorphism [Count of Participants; unit: Participants] — The MTHFR A1298C polymorphism reduces MTHFR enzyme activity; therefore, these patients have higher risk factors for coronary artery disease, acute myocardial infarction, peripheral vascular artery disease, stroke, or venous thromboembolism; having increased basal homocysteine levels or an abnormal methionine-load test (e.g., deficiency of vitamins B12, B6, and folic acid). Population: Some patients had missing genotypes
  Participants
    number analyzed (Participants) | 243 | 244 | 102 | 589
    1298AA | 133 | 120 | 50 | 303
    1298AC | 86 | 105 | 45 | 236
    1298CC | 24 | 19 | 7 | 50
Medications Aspirin [Count of Participants; unit: Participants] | 126 | 137 | 69 | 332
Medications Clopidogrel [Count of Participants; unit: Participants] | 42 | 45 | 24 | 111
Medications Warfarin [Count of Participants; unit: Participants] | 28 | 21 | 13 | 62
Medications Beta-Blocker [Count of Participants; unit: Participants] | 119 | 141 | 70 | 330
ACE-Inhibitor [Count of Participants; unit: Participants] | 94 | 88 | 43 | 225
Statin [Count of Participants; unit: Participants] | 130 | 146 | 69 | 345
Diuretic [Count of Participants; unit: Participants] | 79 | 87 | 28 | 194
Surgical procedure Vascular [Count of Participants; unit: Participants] | 76 | 87 | 53 | 216
Surgical procedure Orthopedic [Count of Participants; unit: Participants] | 88 | 81 | 25 | 194
Surgical procedure ENT [Count of Participants; unit: Participants] | 22 | 20 | 17 | 59
Surgical procedure gyn [Count of Participants; unit: Participants] | 26 | 21 | 8 | 55
Surgical procedure Urology [Count of Participants; unit: Participants] | 22 | 22 | 6 | 50

OUTCOME MEASURES:

1. Primary Outcome: Myocardial Ischemia
Description: Measured by serial troponin and ECG
Time Frame: first 3 postoperative days
Measure: Count of Participants; unit: Participants
Groups:
- B-Vitamin Group: Vitamin B12 and folic acid
  Vitamin B12 and folic acid: 1 mg vitamin B12 IV 5 mg folic acid IV in 100 ml NS infusion
- Standard of Care: Patients did neither receive nitrous oxide nor B-vitmamins
Arm/Group | B-Vitamin Group | Comparator | Standard of Care
Number analyzed (Participants) | 250 | 250 | 125
Participants
  Cardiac troponin elevation | 33 | 34 | 17
  No Cardiac troponin elevation | 217 | 216 | 108

2. Secondary Outcome: Non-fatal MI
Description: Myocardial Infarction per Third Definition of MI
Time Frame: 30 day postoperative
Measure: Count of Participants; unit: Participants
Groups:
- B-Vitamin Group: Vitamin B12 and folic acid
- Standard of Care: No nitrous oxide No B-vitamins
Arm/Group | B-Vitamin Group | Comparator | Standard of Care
Number analyzed (Participants) | 250 | 250 | 125
Participants | 7 | 15 | 8

ADVERSE EVENTS:
Time Frame: 30 day
Arm/Group | Treatment | Comparator | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/250 | 3/250 | 1/125
Serious Adverse Events (participants affected / at risk) | 0/250 | 3/250 | 1/125
Other Adverse Events (participants affected / at risk) | 39/250 | 61/250 | 27/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=250) | Comparator (N=250) | Standard of Care (N=125)
Death (Cardiac disorders) | 0 | 3 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=250) | Comparator (N=250) | Standard of Care (N=125)
Readmission (General disorders) | 9 | 23 | 13
Wound Infection (Infections and infestations) | 15 | 18 | 5
Any Pulmonary (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Cardiovascular (Cardiac disorders) | 5 | 11 | 1
Renal (Renal and urinary disorders) | 0 | 0 | 1
Bleeding (Blood and lymphatic system disorders) | 4 | 2 | 2
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Deep venous thrombosis (Vascular disorders) | 2 | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes